CLINICAL TRIAL: NCT01440283
Title: A Phase II Study of Intensity Modulated Radiation Therapy (IMRT) in High Risk Abdominal Neuroblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBIMRT
Record Dates: First submitted 2011-09-20; First posted 2011-09-26 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2015-11

CONDITIONS: Abdominal Neuroblastoma
Keywords: Neuroblastoma; Radiation Therapy
MeSH Terms: conditions — Neuroblastoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients with high-risk abdominal neuroblastoma who receive any high-risk neuroblastoma treatment regimen will be eligible to enroll prior to surgical resection of the primary tumor. Following implantation of fiducial markers within the tumor bed and autologous hematopoietic rescue, patients will begin the planning process for abdominal irradiation.
  Interventions: Intensity Modulated Radiation Therapy (IMRT)
  Interventions: Radiation: Intensity Modulated Radiation Therapy (IMRT)

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy (IMRT) — IMRT delivery will follow current conventional volume-targeting guidelines, however, appropriate application within the abdomen will be determined by ascertaining intra-abdominal organ motion and the potential for reducing normal tissue dose, while simultaneously increasing dose delivered to target tissues, particularly when dose escalation for gross residual disease is required. Concurrent neuro-hormonal tests, cytokine analyses, functional and morphologic imaging will generate novel data describing the acute and chronic effects of radiotherapy within the abdomen.
  Other Names: IMRT

SUMMARY:
High risk neuroblastoma (NB) is an aggressive, prevalent non-brain cancer derived from nerve cells of the body. It mostly affects infants, and more children die from this tumor each year than are cured. Standard therapy includes a combination of chemotherapy, surgery, bone marrow transplant, radiation and immunotherapy. NB is very sensitive to radiation, but due to it's aggressive spread pattern, radiation use is currently limited by toxicity. This study seeks to improve delivery of radiation to reduce toxicity by quantifying outcomes, and measuring differences in renal toxicity and organ motion so that radiation can be focused more effectively against tumor while sparing normal tissues and reducing side-effects.

DETAILED DESCRIPTION:
Patients with high-risk abdominal neuroblastoma who receive any high-risk neuroblastoma treatment regimen will be eligible to enroll prior to surgical resection of the primary tumor. Following implantation of fiducial markers within the tumor bed and autologous hematopoietic rescue, patients will begin the planning process for abdominal irradiation; this requires multiple baseline studies, including computed tomography (CT), magnetic resonance imaging (MRI), renal scintigraphy, and bloodwork. Most of these tests will be repeated on a varying schedule over the five year follow-up period of the protocol, in order to evaluate the impact of conformal radiotherapy on intra-abdominal tissues.

Intensity modulated radiation therapy (IMRT) delivery will follow current conventional volume-targeting guidelines, however, appropriate application within the abdomen will be determined by ascertaining intra-abdominal organ motion and the potential for reducing normal tissue dose, while simultaneously increasing dose delivered to target tissues, particularly when dose escalation for gross residual disease is required. Concurrent neuro-hormonal tests, cytokine analyses, functional and morphologic imaging will generate novel data describing the acute and chronic effects of radiotherapy within the abdomen.

NOTE: This study is currently closed to accrual, however, it is expected to re-open to accrual later in 2015.

ELIGIBILITY:
Inclusion Criteria:

* Mucositis ≤ Grade 2
* Patient stable on room air
* Albumin > 3 g/dL without albumin infusions for 1 week
* Serum creatinine should be < 1.5 x normal for age
* Lansky score >60
* Risk Strata Eligibility: Patients between 6 months and 18 years of age with newly diagnosed abdominal primary, high-risk neuroblastoma defined as one of the following:

  * International agreement on staging (INSS) stage 2a or 2b with N-myc (MYCN) amplification (greater than four-fold increase in (MYCN) signals as compared to reference signals), regardless of age or additional biologic features
  * INSS stage 3 with either MYCN amplification (greater than four-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features, or for age > 18 months with unfavorable pathology, regardless of MYCN status
  * INSS stage 4 with MYCN amplification (greater than four-fold increase in MYCN signals as compared to reference signals), regardless of age or additional biologic features, or for age >18 months with unfavorable pathology, regardless of MYCN status
  * INSS stage 4S with MYCN amplification (greater than four-fold increase in MYCN signals as compared to reference signals), regardless of additional biologic features
* Exceptional Cases Still Considered Eligible:

  * Prior palliative radiotherapy if not related to the primary site, however, children receiving definitive radiotherapy as a part of the pre-enrollment regimen are ineligible. Prior treatment regimen must follow the guidelines of an applicable high-risk neuroblastoma regimen. Slight variations from this timeframe are acceptable based on recovery of blood counts or other concerns left to the discretion of the treating radiation oncologist.
  * Patients receiving surgical management elsewhere are still considered eligible to enroll on protocol therapy for assessment of the primary local control objective, renal motion and toxicity assessment. Target motion objectives may be excluded from the analysis of these patients.

Exclusion Criteria

* Patients who have received prior definitive radiotherapy at or adjacent to the primary abdominal tumor bed.
* Patients who are unable to cooperate with acquisition of 4-dimensional computed tomography (4DCT), computed tomography (CT) or magnetic resonance imaging- (MRI)-based imaging procedures.
* Patients with known brain metastases.
* Any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
* Pregnant women.
* Mediastinal primary tumors.
* Patients receiving surgery elsewhere, or at St. Jude within 3 months prior to study activation, are excluded from assessment of target and motion objectives. However they are still eligible to enroll for assessment of the primary objective, renal motion and toxicity.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ho Hua, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fourteen participants were enrolled on the study between September 2011 and July 2013.
Groups:
- Treatment: Patients with high-risk abdominal neuroblastoma who receive any high-risk neuroblastoma treatment regimen were eligible to enroll prior to surgical resection of the primary tumor. Following implantation of fiducial markers within the tumor bed and autologous hematopoietic rescue, patients began the planning process for abdominal irradiation.
  Intensity Modulated Radiation Therapy (IMRT) delivery followed current conventional volume-targeting guidelines, however, appropriate application within the abdomen was determined by ascertaining intra-abdominal organ motion and the potential for reducing normal tissue dose, while simultaneously increasing dose delivered to target tissues, particularly when dose escalation for gross residual disease was required.
Period: Overall Study
Arm/Group | Treatment
Started | 14
Completed | 4
Not Completed | 10
Not completed — Death | 3
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.9 (3.1)
Age, Continuous [Median (Full Range); unit: years] | 4.1 [0.9 to 10.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Failed to Reach Local-regional Control
Description: Measured from start of radiation therapy to date of local-regional failure or last follow-up.
Time Frame: 2 years after last patient enrollment
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 14
percentage of participants | 0

2. Primary Outcome: Pattern of Local-regional Failure.
Description: Categorical measurements of local-regional failure.
Time Frame: 2 years after last patient enrollment
Population: There was no local-regional failure noted (please see outcome #1), therefore, no pattern of failure could be determined.
Arm/Group | Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Quantify the Range of Organ Movement During the Breathing Phase Measured by 4-dimensional MRI (4DMRI) and 4DCT.
Description: Normal tissue motion-defining measurements were obtained which can guide future more conformal therapeutic regimens incorporating smaller volumes of uninvolved tissue. Participants underwent CT simulation and 4D-CT acquisition as well as real-time dynamic 4D MRI prior to the start of radiation therapy (RT), and a subsequent repeat 4D-CT was obtained approximately 2 weeks after the start of RT. The imaging position was supine with general anesthesia. Renal edges were marked in a customized graphical interface for each imaging series with the image resolution determining the minimum motion extent. Vectors of renal edge motion were quantified in the anterior-posterior (A-P), medial-lateral (M-L), and superior-inferior (S-I) dimensions. The motion extent derived from the MRI dataset was considered in defining the margins for RT treatment planning.
Time Frame: Baseline and approximately 2 weeks following initiation of irradiation.
Population: Five participants did not receive all scans for motion evaluations and are excluded from the analysis. Age at scan ranges from 8 months to 9.5 years old. The median age was 3.8 years.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Right Kidney: M-L; Right Kidney: A-P; Right Kidney: S-I; Left Kidney: M-L; Left Kidney: A-P; Left Kidney: S-I: Nine participants who underwent all 3 scans.
Arm/Group | Right Kidney: M-L | Right Kidney: A-P | Right Kidney: S-I | Left Kidney: M-L | Left Kidney: A-P | Left Kidney: S-I
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9
mm
  Baseline 4D CT | 0.3 (0.4) | 0.5 (0.5) | 2.6 (1.5) | 0.5 (0.5) | 0.4 (0.4) | 2.2 (1.8)
  Week 2 4D CT | 0.4 (0.3) | 0.4 (0.4) | 2.8 (0.8) | 0.5 (0.3) | 0.5 (0.2) | 2.3 (1.3)
  Baseline MRI | 0.8 (1.0) | 0.5 (0.7) | 2.6 (0.8) | 0.5 (0.7) | 0.3 (0.6) | 2.3 (0.8)

4. Secondary Outcome: Quantify (in mm/cm) the Range of Target Movement During the Breathing Phase Measured by 4DMRI and 4DCT.
Description: Obtain target tissue motion-defining data which can guide future more conformal therapeutic regimens incorporating smaller volumes of uninvolved tissue.
Time Frame: Baseline and approximately 2 weeks following initiation of irradiation.
Population: All participants underwent complete surgery prior to RT, therefore, no visible tumor tissue target was available for movement measurements.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the initiation of radiation therapy until completion of study, removal from study, or disease recurrence, up to 2 years after the last participant enrollment.
Description: The therapy delivered on protocol was standard of care (standard indications for radiation and standard radiation doses) and was not expected to generate unexpected toxicities related to abdominal radiation.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=14)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=14)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 8 (21)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (2)
Platelet count decreased (Blood and lymphatic system disorders) | 5 (11)
White blood cell decreased (Blood and lymphatic system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was closed to accrual in January 2014 due to the principal investigator leaving St. Jude. It was expected to re-open to accrual, however, in September 2015, the decision was made to permanently close the trial to participant enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes